CLINICAL TRIAL: NCT01992965
Title: Effect of Real-time Continuous Glucose Monitoring on Glucose Control and Outcomes of Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kang Yan (Other)
Responsible Party: Sponsor-Investigator, Kang Yan, Director of Intensive Care Unit, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CGM-ky0521
Record Dates: First submitted 2013-11-13; First posted 2013-11-25 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Hyperglycemia
Keywords: continuous glucose monitoring；; critically ill;
MeSH Terms: conditions — Hyperglycemia; Critical Illness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous Glucose Monitoring Group (Experimental): Continuous Glucose Monitoring Group:
  Different methods of blood glucose monitoring between groups, and this group will use real-time continuous glucose monitoring system with alarm limits（high and low limit is 10 mmol/L and 8 mmil/L , respectively ) up to five days for glucose control, the target mean glucose level is between 8 and 10 mmol/L.
  Interventions: Other: Different methods of blood glucose monitoring between groups
- Conventional Group (Active Comparator): Conventional Group：
  Different methods of blood glucose monitoring between groups, and this group will use finger prick blood glucose measurements for glucose control with the same target mean glucose level of 8 -10 mmol/L. Patients also wear real-time continuous glucose monitoring system to collect glucose measurements. The values of real-time continuous glucose monitoring system are blinded to investigator and patients.
  Interventions: Other: Different methods of blood glucose monitoring between groups

INTERVENTIONS:
Other: Different methods of blood glucose monitoring between groups — Finger prick blood glucose in conventional group versus real-time continuous glucose monitoring system of continuous glucose monitoring group

SUMMARY:
The purpose of the study is to evaluate the effect of real-time continuous glucose monitoring system on glucose control and outcomes of critically ill patients.

DETAILED DESCRIPTION:
Real-time continuous glucose monitoring system has shown great accuracy and feasibility in critically ill patients. However, its impact on glucose control and outcomes has nearly unknown. Thus, Investigators designed this study to evaluate the effect of real-time continuous glucose monitoring system on glucose control and outcomes of critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old male or female;

  * Expected ICU stays longer than 72 hours;

    * Glucose level more than 8 mmol/L when enrolls in the ICU;

      * Patients or their legal surrogates have signed the informed consent.

Exclusion Criteria:

* Pregnant or lactating women;

  * ICU stays less than 72 hours;

    * Usage of real-time continuous glucose monitoring system is considered as a contraindication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Glycemic Control Measures including: Percentage of target blood glucose levels (defined as between 8mmol/L and 10mmol/L); Time of hyperglycemia (defined as >10mmol/L); Hypoglycemia rate (defined as < 2.2mmol/L); Glucose lability index | Glycemic control measures will be assessed up to five days.

SECONDARY OUTCOMES:
Prognosis Measures including: Duration of mechanical ventilation；Time of ICU stay; Time of hospital stay; 28 days - mortality rate | All the participants will be followed for the duration of hospital stay or 28 days.
Cost | Cost associated with glucose monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Yan Kang, MD, Study Director — West China Hospital
Locations (1):
- Intensive care unit of West China Hospital, Chengdu, Sichuan, China